CLINICAL TRIAL: NCT02474888
Title: Pharmacokinetic Study of Rituximab Induction Regimen in ANCA-associated Vasculitis : a Predictive Factor of Clinical Outcome? (MONITUX)
Brief Title: Pharmacokinetic Study of Rituximab Induction Regimen in ANCA-associated Vasculitis
Acronym: MONITUX
Status: Terminated | Type: Observational
Why Stopped: failure of recruit
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Theradiag (Other)
Responsible Party: Sponsor
Other Study IDs: 1508058; 2015-001807-29 (EudraCT Number)
Record Dates: First submitted 2015-06-10; First posted 2015-06-18 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Granulomatosis, Wegener's; Microscopic Polyangiitis
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood specimen for serum rituximab level and serum anti-rituximab level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rituximab: a classical induction regimen with rituximab (decision taken before inclusion), implying an infusion of 375mg/m² per week, for 4 consecutive weeks (from week -3 until week 0) with blood specimen.
  Interventions: Other: blood specimen

INTERVENTIONS:
Other: blood specimen — blood specimen for serum rituximab level and serum anti-rituximab level at M1 and M3 after stop of induction rituximab treatment

SUMMARY:
The aim of the investigators' study is to evaluate whether monitoring serum rituximab levels could be an interesting tool in the follow-up of ANCA-associated vasculitis patients.

All consecutive patients, hospitalized for a new diagnosis of ANCA-associated vasculitis or the relapse of a known ANCA-associated vasculitis, in which the decision to start an induction regimen with rituximab has been taken, will be included.

Serum rituximab levels (along with serum anti-rituximab antibodies levels) will be determined (at M+1 and M+3) and the correlation with clinical outcome at M+6 will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Granulomatosis with polyangiitis or microscopic polyangiitis (according to Chapel Hill criterions), with or without detectable ANCA
* Decision taken to start an induction regimen with rituximab
* Informed and having signed the study consent form
* If of child-bearing potential, female patients will have use an effective method of contraception during RTX (rituximab) treatment and in the 12 months following RTX treatment stop
* no-breast-feeding during RTX treatment and in the 12 months following RTX treatment stop

Exclusion Criteria:

* Other primary or secondary systemic vasculitis
* Incapacity or refusal to sign the informed consent form
* Incapacity or refusal to adhere to treatment or perform the follow-up examinations required by the study
* Allergy, documented hypersensitivity or contraindication to the medications used in the present study (corticosteroids, rituximab)
* severe active infection
* Patient with severe heart failure (stage NYHA IV) or any other unstable heart disease Pregnancy, except for cases where the expected benefit oj treatment seems to surpass the potential risks
* Patients with active hepatitis B
* Any live vaccine within four weeks prior to the first infusion of RTX

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Granulomatosis with polyangiitis or microscopic polyangiitis (according to Chapel Hill criterions), with or without detectable ANCA
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
serum rituximab levels | 1 month after stop of rituximab induction regimen
  rituximab level comparison between number of non-responders and number of responders after rituximab induction regimen. The number of non-responders is defined by a Birmingham Vascularitis Activity score > 0, 6 months after stop of induction regimen

SECONDARY OUTCOMES:
serum rituximab levels | 3 months after stop of rituximab induction regimen
  rituximab level comparison between number of non-responders and number of responders after rituximab induction regimen. The number of non-responders is defined by a Birmingham Vascularitis Activity score > 0 six months after stop of induction regimen
serum rituximab levels | 6 months after stop of rituximab induction regimen
  rituximab level comparison between number of non-responders and number of responders after rituximab induction regimen. The number of non-responders is defined by a Birmingham Vascularitis Activity score > 0 six months after stop of induction regimen
serum anti-rituximab antibodies | 1 month after stop of rituximab induction regimen
  serum anti-rituximab antibodies level comparison between number of non-responders and number of responders after rituximab induction regimen. The number of non-responders is defined by a Birmingham Vascularitis Activity score > 0 six months after stop of induction regimen
serum anti-rituximab antibodies | 3 months after stop of rituximab induction regimen
  serum anti-rituximab antibodies level comparison between number of non-responders and number of responders after rituximab induction regimen. The number of non-responders is defined by a Birmingham Vascularitis Activity score > 0 six months after stop of induction regimen
serum anti-rituximab antibodies | 6 months after stop of rituximab induction regimen
  serum anti-rituximab antibodies level comparison between number of non-responders and number of responders after rituximab induction regimen. The number of non-responders is defined by a Birmingham Vascularitis Activity score > 0 six months after stop of induction regimen
Serum B lymphocytes (CD19+ cells) levels | 1 month after stop of rituximab induction regimen
  Serum B lymphocytes (CD19+ cells) levels comparison between number of non-responders and number of responders after rituximab induction regimen. The number of non-responders is defined by a Birmingham Vascularitis Activity score > 0 six months after stop of induction regimen
Serum B lymphocytes (CD19+ cells) levels | 3 months after stop of rituximab induction regimen
  Serum B lymphocytes (CD19+ cells) levels comparison between number of non-responders and number of responders after rituximab induction regimen. The number of non-responders is defined by a Birmingham Vascularitis Activity score > 0 six months after stop of induction regimen
Serum B lymphocytes (CD19+ cells) levels | 6 months after stop of rituximab induction regimen
  Serum B lymphocytes (CD19+ cells) levels comparison between number of non-responders and number of responders after rituximab induction regimen. The number of non-responders is defined by a Birmingham Vascularitis Activity score > 0 six months after stop of induction regimen
patient number with adverse event | from start of induction rituximab regimen until six monthes after stop of induction regimen
  frequency and nature of rituximab-attributed adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Pascal CATHEBRAS, PHD, Principal Investigator — CHU SAINT-ETIENNE
Locations (4):
- France (4):
  - Hôpital Edouard Herriot, Lyon
  - Hôpital de la Croix Rousse, Lyon
  - CH Lyon Sud, Pierre-Bénite
  - CHU Saint-Etienne, Saint-Etienne